CLINICAL TRIAL: NCT00870688
Title: Non Interventional Trial of Valproate Sustained Release Minitablets Once Daily in the Evening
Brief Title: Valproate Sustained Release Minitablets (Orfiril(R) Long) Once Daily in the Evening
Status: Completed | Type: Observational
Sponsor: Desitin Arzneimittel GmbH (Industry)
Responsible Party: Karin Lohmueller, Desitin Arzneimittel GmbH
Other Study IDs: VPA 044/K
Record Dates: First submitted 2009-01-09; First posted 2009-03-27 (Estimated); Results first posted 2009-03-27 (Estimated); Last update posted 2009-05-20 (Estimated); Status verified 2009-02

CONDITIONS: Epilepsy
Keywords: valproate; epilepsy; compliance; sustained released minitablet; Orfiril long
MeSH Terms: conditions — Epilepsy; Patient Compliance | interventions — Valproic Acid

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: epilepsy patients
  Interventions: Drug: sodium valproate

INTERVENTIONS:
Drug: sodium valproate — valproate sustained release minitablets, once daily.
  Other Names: Orfiril (R) long

SUMMARY:
Valproate is the first line therapy in primary generalized seizures. The applied drug contains sodium valproate in sustained release minitablets. As a multiple unit dosage form these can be easily swallowed and taken independent from meals.

A simple dosage scheme like valproate sustained release minitablets once daily in the evening should improve the compliance and likely the seizure situation of the patients. The data of this non interventional trial were directly extracted from the physician's electronic patient database. The observational period was 7 weeks compared to a retrospective period 7 weeks before start of the study.

ELIGIBILITY:
Inclusion Criteria:

* age of 12 years and above
* epilepsy patients
* indication to initiation / conversion to valproate sustained release minitablets once daily

Exclusion Criteria:

* contraindication to valproate use
* no indication for conversion to valproate sustained release minitablets once daily

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: community sample outpatients
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2005-01; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In total 82 patients were included in this trial. The patients were naive or changed from another antiepileptic or valproate preparation to valproate sustained release minitablets once daily in the evening.
Groups:
- Sodium Valproate: Epilepsy patients receive valproate sustained release minitablets, once daily.
Period: Overall Study
Arm/Group | Sodium Valproate
Started | 82
Completed | 78
Not Completed | 4
Not completed — Lost to Follow-up | 2
Not completed — Death, Unrelated | 1
Not completed — Granules in the Stools | 1

BASELINE CHARACTERISTICS:
Arm/Group | Sodium Valproate
Number analyzed (Participants) | 82
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 61
  >=65 years | 20
Age Continuous [Mean (Standard Deviation); unit: years] | 45.9 (23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43
  Male | 39

OUTCOME MEASURES:

1. Primary Outcome: Change in Number of Seizures After Conversion To Valproate Retard Minitablets Once Daily
Time Frame: 7 weeks
Reporting Status: Not Posted
Measure: unit: number of seizures

2. Secondary Outcome: Data About Efficacy, Safety and Compliance
Time Frame: 7 weeks
Reporting Status: Not Posted

3. Primary Outcome: Number of Seizures Within 7 Weeks
Time Frame: 7 weeks
Measure: Mean (Standard Deviation); unit: seizures
Arm/Group | Sodium Valproate
Number analyzed (Participants) | 82
seizures | 1.6 (2.9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No